CLINICAL TRIAL: NCT04372394
Title: A Phase 1, Two Period Crossover Study to Assess the Effect of a High Fat Meal on the Pharmacokinetics of Surufatinib in Healthy Subjects
Brief Title: A Study to Assess the Effect of a High Fat Meal on Surufatinib in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-012-00US1
Record Dates: First submitted 2020-04-14; First posted 2020-05-04 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2020-07

CONDITIONS: Healthy
MeSH Terms: interventions — surufatinib

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to 1 of the 2 possible treatment sequences as follows:
  * Fed/Fasted: surufatinib with food on Day 1 and surufatinib without food on Day 8
  * Fasting/Fed: surufatinib without food on Day 1 and surufatinib with food on Day 8
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fed/Fasted (Experimental): surufatinib with food on Day 1 and surufatinib without food on Day 8
  Interventions: Drug: surufatinib
- Fasted/Fed (Experimental): surufatinib without food on Day 1 and surufatinib with food on Day 8
  Interventions: Drug: surufatinib

INTERVENTIONS:
Drug: surufatinib — Surufatinib: 300 mg as a single dose on Days 1 and 8 with or without food

SUMMARY:
This study will be a 2-period study conducted with 26 healthy male or female subjects. Subjects will be randomly assigned to either receive a single dose of surufatinib with food in period 1, then without food in period 2, or vice-versa.

DETAILED DESCRIPTION:
This study will be a single center, open label, randomized crossover, 2-period study conducted with 26 healthy male or female subjects. Subjects will be randomly assigned to 1 of the 2 possible treatment sequences as follows:

* Fed/Fasted: surufatinib with food on Day 1 and surufatinib without food on Day 8
* Fasting/Fed: surufatinib without food on Day 1 and surufatinib with food on Day 8

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, healthy male or female between the ages of 18 and 55 years old inclusive).
* Body mass index (BMI) > 18 and ≤ 29 kg/m2.
* Females must be of non-childbearing potential, or of childbearing potential and agree to use a medically acceptable method of contraception.
* Males who have not had a successful vasectomy and are partners of women of childbearing potential must use, or their partners must use, a highly effective method of contraception starting for at least one menstrual cycle prior to and throughout the entire study period, and for 2 weeks after the last dose of study drug. Those with partners using hormonal contraceptives must also use an additional approved method of contraception. No sperm donation is allowed during the study period and for 90 days after study drug discontinuation.

Exclusion Criteria:

* Evidence of clinically significant cardiovascular, hepatic, GI, renal, respiratory, endocrine, hematological, neurological, or psychiatric disease or abnormalities or had a known history of any GI surgery or cholecystectomy.
* Clinically significant illness within 8 weeks or had a clinically significant infection within 4 weeks prior to the first dose.
* Known food allergy to any content of the standard meal to be used in this study.
* Clinically significant deviation from normal in the physical examination, vital signs, or clinical laboratory determinations.
* Systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg.
* The subject has a clinically significant ECG abnormality, or had a family history of prolonged QTc syndrome or sudden death.
* A history of smoking or use of nicotine-containing substances within the previous 2 months.
* A history of drug or alcohol misuse in the previous 6 months.
* Has been diagnosed with acquired immune deficiency syndrome (AIDS) or are positive for human immunodeficiency virus (HIV), Hepatitis B virus (HBV), or Hepatitis C virus (HCV).
* Has participated in a clinical trial of other drug before screening, and the time since the last use of other study drug is less than 5 times the half- life or 4 weeks, whichever is longer, or the subject is currently enrolled in another clinical trial.
* Has received blood or blood products within 4 weeks, or donated blood or blood products within 8 weeks.
* Has used any over-the-counter (OTC) medications or prescription drugs within 2 weeks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
AUC (0-t) of Surufatinib | Up to Day 15
  Pharmacokinetics of surufatinib by assessment of area under the plasma concentration time curve from zero to the last measurable concentration
AUC of Surufatinib | Up to Day 15
  Pharmacokinetics of surufatinib by assessment of area under the plasma concentration curve from zero extrapolated to infinity
Cmax of Surufatinib | Up to Day 15
  Pharmacokinetics of Surufatinib by assessment of maximum plasma Surufatinib concentration

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events as assessed by CTCAE v5.0 | Up to Day 15
  To evaluate the safety, in healthy subjects, of a single dose of surufatinib administered with and without food

CONTACTS AND LOCATIONS:
Overall Officials: Jeanelle Kam, MD, Principal Investigator — Covance Clinical Research Unit
Locations (1):
- Covance Clinical Research Unit, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No